CLINICAL TRIAL: NCT01025739
Title: Phase II Study of Evaluation of the Safety and Effectiveness of Tailored Transoral Incisionless Fundoplication (TIF) Using EsophyX for the Treatment of GERD
Brief Title: Evaluation of the Safety and Effectiveness of Tailored Transoral Incisionless Fundoplication (TIF) Using EsophyX for the Treatment of GERD
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No funding source for device purchasing
Sponsor: University of Alberta (Other)
Collaborators: AHS Cancer Control Alberta (Other)
Responsible Party: Principal Investigator, Daniel Birch, MSc, MD, FRCSC, FACS, University of Alberta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00004475
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: Gastroesophageal Reflux Disease (GERD); EsophyX
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: EsophyX™ system with SerosaFuse fasteners — The EsophyX™ system with SerosaFuse fasteners (EndoGastric Solutions, Redmond, WA, USA) was designed to reconstruct the gastroesophageal junction through anterior partial fundoplication with tailored delivery of multiple fasteners during a single-device insertion.

SUMMARY:
Objectives of the Study:

The primary objective of this study is to evaluate the relative merits, safety and effectiveness of the tailored TIF2 procedure in treating GERD patients who have persistent GERD symptoms despite PPI therapy.

The secondary objective of the study is to evaluate the effectiveness of the tailored TIF procedure in restoring the antireflux barrier and eliminating GE reflux.

Type of Study:

Prospective, non-randomized, uncontrolled Study Duration 12 months Number of Patients 20

Inclusion Criteria:

Age 18-70 years, on daily PPIs for > 6 months, persistent GERD symptoms despite PPI therapy, anatomic disruption of the gastroesophageal valve to a Hill Grade II-III, evidence of one of the following while on PPI therapy: (1) erosive esophagitis (erosions or ulcerations during endoscopy); (2) abnormal ambulatory pH study; or (3) biopsy confirmed changes characteristic of reflux esophagitis; acceptable esophageal motility (by either manometry or video esophagogram), hiatal hernia no larger than 2 cm, patient willing to cooperate with post-operative dietary recommendations and assessment tests, signed informed consent

Exclusion Criteria:

BMI > 40, hiatal hernia > 2 cm, esophagitis grade D, esophageal ulcer, fixed esophageal stricture, gastric motility disorders, previous splenectomy, pregnancy (female), immunosuppression, ASA > 2, portal hypertension and/or varices, history of previous resective gastric or esophageal surgery, cervical spine fusion, Zenker's diverticulum, esophageal epiphrenic diverticulum, achalasia, scleroderma or dermatomyositis, eosinophilic esophagitis, or cirrhosis, active gastro-duodenal ulcer disease, gastric outlet obstruction or stenosis, gastroparesis or delayed gastric emptying, coagulation disorders

Interventions:

Treatment: Tailored transoral incisionless fundoplication (TIF2) using EsophyX system with SerosaFuse fasteners (EndoGastric Solutions, Inc., Redmond, WA, USA)

Evaluation Criteria:

Primary Outcome Measure 24 hour pH impedance study: change in Johnson DeMeester scores; GERD-HRQOL scores Secondary Outcome Measures PPI usage, GERD symptoms at 6 and 12 months vs. baseline off PPI's, total number of reflux episodes, and Symptom Association Probability while off PPI.

Safety: Adverse events will be mapped to standard terms and reported.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* On daily PPIs for > 6 months
* Persistent GERD symptoms despite PPI therapy
* Anatomic disruption of the gastroesophageal valve to a Hill Grade II-III
* Evidence of one of the following while on PPI therapy:

  * Erosive esophagitis (erosions or ulcerations during endoscopy)
  * Abnormal ambulatory pH study
  * Biopsy confirmed changes characteristic of reflux esophagitis
* Acceptable esophageal motility (by either manometry or video esophagogram)
* Hiatal hernia no larger than 2 cm
* Patient willing to cooperate with post-operative dietary recommendations and assessment tests
* Signed informed consent

Exclusion Criteria:

* BMI > 40
* Hiatal hernia > 2 cm
* Esophagitis grade D
* Esophageal ulcer
* Esophageal stricture
* Esophageal motility disorder
* Prior splenectomy
* Pregnancy or plans for pregnancy in the next 12 months (in females)
* Immunosuppression
* ASA > 2
* Portal hypertension and/or varices
* History of previous resective gastric or esophageal surgery, cervical spine fusion, Zenker's diverticulum, esophageal epiphrenic diverticulum, achalasia, scleroderma or dermatomyositis, eosinophilic esophagitis, or cirrhosis
* Active gastro-duodenal ulcer disease
* Gastric outlet obstruction or stenosis
* Gastroparesis or delayed gastric emptying confirmed by solid-phase gastric emptying study if patient complains of postprandial satiety during assessment
* Coagulation disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
24 hour pH impedance study: change in Johnson DeMeester scores; GERD-HRQOL scores | 1, 3, 6, 12 month

SECONDARY OUTCOMES:
PPI usage, GERD symptoms at 6 and 12 months vs. baseline off PPI's, total number of reflux episodes, and Symptom Association Probability while off PPI. Safety: Adverse events will be mapped to standard terms and reported. | 1 day; 1 week; 1, 3, 6, 12 month

CONTACTS AND LOCATIONS:
Locations (1):
- CAMIS, Royal Alexandra Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] El-Serag HB. Time trends of gastroesophageal reflux disease: a systematic review. Clin Gastroenterol Hepatol. 2007 Jan;5(1):17-26. doi: 10.1016/j.cgh.2006.09.016. Epub 2006 Dec 4. PMID 17142109
- [Background] Lundell L. Surgery of gastroesophageal reflux disease: a competitive or complementary procedure? Dig Dis. 2004;22(2):161-70. doi: 10.1159/000080315. PMID 15383757
- [Background] Metz DC. Managing gastroesophageal reflux disease for the lifetime of the patient: evaluating the long-term options. Am J Med. 2004 Sep 6;117 Suppl 5A:49S-55S. doi: 10.1016/j.amjmed.2004.07.009. PMID 15478853
- [Background] Moayyedi P, Talley NJ. Gastro-oesophageal reflux disease. Lancet. 2006 Jun 24;367(9528):2086-100. doi: 10.1016/S0140-6736(06)68932-0. PMID 16798392
- [Background] Nandurkar S, Talley NJ. Epidemiology and natural history of reflux disease. Baillieres Best Pract Res Clin Gastroenterol. 2000 Oct;14(5):743-57. doi: 10.1053/bega.2000.0122. PMID 11003807
- [Background] Smout AJ. The patient with GORD and chronically recurrent problems. Best Pract Res Clin Gastroenterol. 2007;21(3):365-78. doi: 10.1016/j.bpg.2007.01.007. PMID 17544105
- [Background] Stylopoulos N, Rattner DW. The history of hiatal hernia surgery: from Bowditch to laparoscopy. Ann Surg. 2005 Jan;241(1):185-93. doi: 10.1097/01.sla.0000149430.83220.7f. PMID 15622007
- [Background] Jones MP, Sloan SS, Rabine JC, Ebert CC, Huang CF, Kahrilas PJ. Hiatal hernia size is the dominant determinant of esophagitis presence and severity in gastroesophageal reflux disease. Am J Gastroenterol. 2001 Jun;96(6):1711-7. doi: 10.1111/j.1572-0241.2001.03926.x. PMID 11419819
- [Background] Mittal RK. Hiatal hernia: myth or reality? Am J Med. 1997 Nov 24;103(5A):33S-39S. doi: 10.1016/s0002-9343(97)00318-5. No abstract available. PMID 9422620
- [Background] Mittal RK. Hiatal hernia and gastroesophageal reflux: another attempt to resolve the controversy. Gastroenterology. 1993 Sep;105(3):941-3. doi: 10.1016/0016-5085(93)90917-2. No abstract available. PMID 8359662
- [Background] Moss SF, Kidd M, Modlin IM. The status of the hiatus: the role of hernia in gastroesophageal reflux disease. J Clin Gastroenterol 2007;41:S144-S153
- [Background] Rydberg L, Ruth M, Lundell L. Mechanism of action of antireflux procedures. Br J Surg. 1999 Mar;86(3):405-10. doi: 10.1046/j.1365-2168.1999.01025.x. PMID 10201789
- [Background] Ahroni JH, Montgomery KF, Watkins BM. Laparoscopic adjustable gastric banding: weight loss, co-morbidities, medication usage and quality of life at one year. Obes Surg. 2005 May;15(5):641-7. doi: 10.1381/0960892053923716. PMID 15946454
- [Background] Cadiere GB, Rajan A, Rqibate M, Germay O, Dapri G, Himpens J, Gawlicka AK. Endoluminal fundoplication (ELF)--evolution of EsophyX, a new surgical device for transoral surgery. Minim Invasive Ther Allied Technol. 2006;15(6):348-55. doi: 10.1080/13645700601040024. PMID 17190659
- [Background] Jobe BA, O'Rourke RW, McMahon BP, Gravesen F, Lorenzo C, Hunter JG, Bronner M, Kraemer SJ. Transoral endoscopic fundoplication in the treatment of gastroesophageal reflux disease: the anatomic and physiologic basis for reconstruction of the esophagogastric junction using a novel device. Ann Surg. 2008 Jul;248(1):69-76. doi: 10.1097/SLA.0b013e31817c9630. PMID 18580209
- [Background] Cadiere GB, Rajan A, Germay O, Himpens J. Endoluminal fundoplication by a transoral device for the treatment of GERD: A feasibility study. Surg Endosc. 2008 Feb;22(2):333-42. doi: 10.1007/s00464-007-9618-9. Epub 2007 Dec 11. PMID 18071818
- [Background] Cadiere GB, Buset M, Muls V, Rajan A, Rosch T, Eckardt AJ, Weerts J, Bastens B, Costamagna G, Marchese M, Louis H, Mana F, Sermon F, Gawlicka AK, Daniel MA, Deviere J. Antireflux transoral incisionless fundoplication using EsophyX: 12-month results of a prospective multicenter study. World J Surg. 2008 Aug;32(8):1676-88. doi: 10.1007/s00268-008-9594-9. PMID 18443855
- [Background] Huber-Lang M, Henne-Bruns D, Schmitz B, Wuerl P. Esophageal perforation: principles of diagnosis and surgical management. Surg Today. 2006;36(4):332-40. doi: 10.1007/s00595-005-3158-5. PMID 16554990
- [Background] Bouvy ND, Witteman BPL, Jobe BA, Lorenzo C, Kraemer SJM, Gawlicka AK, McMahon B, Gravesen FH, Masclee A, Hameeteman W, Koek GH, Perry K. Tailored reconstruction of the esophagogastric junction using transoral incisionless fundoplication: a feasibility study. Surg Endosc 2008
- [Background] Witteman BP, Strijkers R, de Vries E, Toemen L, Conchillo JM, Hameeteman W, Dagnelie PC, Koek GH, Bouvy ND. Transoral incisionless fundoplication for treatment of gastroesophageal reflux disease in clinical practice. Surg Endosc. 2012 Nov;26(11):3307-15. doi: 10.1007/s00464-012-2324-2. Epub 2012 May 31. PMID 22648098
- [Background] Bouvy ND, Witteman BPL, de Vries E, van Dam R, Greve JW, Gawlicka AK, Masclee A, Hameeteman W, Koek GH. EsophyX transoral incisionless fundoplication for the treatment of GERD in clinical practice. Gastrointest Endosc 2008
- [Background] Lundell LR, Dent J, Bennett JR, Blum AL, Armstrong D, Galmiche JP, Johnson F, Hongo M, Richter JE, Spechler SJ, Tytgat GN, Wallin L. Endoscopic assessment of oesophagitis: clinical and functional correlates and further validation of the Los Angeles classification. Gut. 1999 Aug;45(2):172-80. doi: 10.1136/gut.45.2.172. PMID 10403727
- [Background] Jobe BA, Kahrilas PJ, Vernon AH, Sandone C, Gopal DV, Swanstrom LL, Aye RW, Hill LD, Hunter JG. Endoscopic appraisal of the gastroesophageal valve after antireflux surgery. Am J Gastroenterol. 2004 Feb;99(2):233-43. doi: 10.1111/j.1572-0241.2004.04042.x. PMID 15046210
- [Background] Hill LD, Kozarek RA, Kraemer SJ, Aye RW, Mercer CD, Low DE, Pope CE 2nd. The gastroesophageal flap valve: in vitro and in vivo observations. Gastrointest Endosc. 1996 Nov;44(5):541-7. doi: 10.1016/s0016-5107(96)70006-8. PMID 8934159